CLINICAL TRIAL: NCT02418689
Title: A Prospective, Open-label, Single-arm, Multi-Center, Phase II Trial of NOV120101 in Patients With HER2-overexpressed Recurrent Stage IV Breast Cancer Who Have Received at Least 2 Prior HER2-directed Regimens
Brief Title: Poziotinib in Patients With HER2+ Recurrent Stage IV BC Who Have Received at Least 2 Prior HER2-directed Regimens
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hanmi Pharmaceutical Company Limited (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NOV120101-203
Record Dates: First submitted 2015-01-19; First posted 2015-04-16 (Estimated); Last update posted 2022-01-20 (Actual); Status verified 2021-03

CONDITIONS: Metastatic Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — HM781-36B

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- NOV120101 (Poziotinib) (Experimental): Single arm study with NOV120101(poziotinib) 12 mg PO once daily for 2 weeks followed by a 1-week drug-free interval
  Interventions: Drug: NOV120101 (Poziotinib)

INTERVENTIONS:
Drug: NOV120101 (Poziotinib) — NOV120101 (Poziotinib) 12 mg PO once daily for 2 weeks followed by a 1-week drug-free interval between cycles until disease progression or unacceptable toxicity development
  Other Names: HM781-36B; Poziotinib

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of novel pan-HER inhibitor, NOV120101 (Poziotinib), in HER2-overexpressed recurrent stage IV breast cancer patients who received at least 2 prior HER2-directed regimens.

DETAILED DESCRIPTION:
To evaluate the efficacy of NOV120101 (Poziotinib) as a therapeutic agent for HER2-overexpressed recurrent stage IV breast cancer, patients who have received at least two prior HER2-directed regimens will be enrolled in this study. Subjects will receive NOV120101 (Poziotinib) 12 mg PO once daily for 2 weeks followed by 1-week drug-free intervals between cycles until disease progression or unacceptable toxicity development. Progression Free Survival (PFS) will be analyzed as the primary endpoint in this trial. Secondary endpoints including PFS rate at 12 weeks, ORR, DCR, OS and TTP will also be analyzed.

ELIGIBILITY:
Inclusion Criteria:

1. Who give agreement to the collection of tumor tissue specimen suitable for biomarker research
2. ECOG performance status ≤ 2
3. Who received following treatments as Taxane-based chemotherapy and at least two HER2-targeted* therapy including Trastuzumab.

   * lapatinib, T-DM1 (trastuzumab emtansine), pertuzumab
4. Adequate hematological, hepatic and renal functions

Exclusion Criteria:

1. Who received NOV120101 prior to participation in this study
2. Patients expected to exhibit hypersensitivity to IP or its components
3. Any other concurrent chemotherapies
4. Concurrent or prior radiotherapy within 4 weeks before study participation. However, patients with additional lesions other than the major lesion who completed and recovered from all treatment-related toxicities after radiotherapy in a limited area as a palliative therapy are allowed to participate in the study
5. History of symptomatic or unstable angina and congestive heart failure; arrhythmia requiring medications; or clinically significant myocardial infarction or other cardiac diseases within 6 months before study participation for which any related-significant risks are expected
6. Patients whose left ventricle ejection fraction (LVEF) is below the institutional lower limit of normal. However, if no lower limit of normal is defined in the site, the lower limit or normal is 50%.
7. Concurrent active hepatic or biliary disease (with exception of Gilbert's syndrome, asymptomatic gallstones, liver metastases or stable chronic liver diseases)
8. History or concurrent ongoing/active infection, or uncontrolled diseases including, but not limited to, psychiatric illness/social situations which may limit the compliance with study procedures
9. Prior chemo-, immuno-, or surgical therapy within 3 weeks, or hormone therapy within 1 week before IP administration
10. History of primary malignancies other than breast cancer.
11. Patients with central nervous system (CNS) metastases.
12. Patients receiving or expected to receive bisphosphonate for prophylactic use without any bone-related diseases during the trial, for the exception of the treatment for bone metastases or osteoporosis initiated prior the IP administration.
13. Clinically significant or recent acute gastrointestinal disorders with diarrhea as a major symptom
14. Who are unstable or with unresolved severe adverse event(s)
15. Pregnancy or breast-feeding
16. Women of childbearing potential or men who are unwilling to use adequate contraception or be abstinent during the trial and for at least 2 months after the end of treatment

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 106 (Actual)
Dates: Start 2015-04 (Actual); Primary Completion 2017-06 (Actual); Study Completion 2021-04 (Actual)

PRIMARY OUTCOMES:
Progression free survival (PFS) | By 12 months after enrollment of the last subject

SECONDARY OUTCOMES:
PFS rate at Week 12 | 12 weeks
Objective Response Rate (ORR) | By 12 months after enrollment of the last subject
  the proportion of patients with complete response (CR) and/or partial response (PR)
Disease Control Rate (DCR) | By 12 months after enrollment of the last subject
  the proportion of patients with CR, PR and/or stable disease (SD)] [Safety Issue?
Duration of Disease Control | By 12 months after enrollment of the last subject
Overall Survival (OS) | By 12 months after enrollment of the last subject
Time To Progression (TTP) | By 12 months after enrollment of the last subject
Time to objective response | By 12 months after enrollment of the last subject
Duration of objective response | By 12 months after enrollment of the last subject

OTHER OUTCOMES:
Population pharmacokinetics (PK) of NOV120101 (Poziotinib) - Ka, CL(clearance), Vd(volume of distribution) | 4 weeks
Number of Participants with Adverse Events as a Measure of Safety and Tolerability | 2 years

CONTACTS AND LOCATIONS:
Locations (7):
- South Korea (7):
  - National Cancer Center, Goyang-si, Gyeonggi-do
  - Seoul National University Bundang Hospital, Seongnam-si, Gyeonggi-do
  - Chungbuk National University Hospital, Cheongju-si, North Chungcheong
  - Samsung Medical Center, Gangnam-gu, Seoul
  - Seoul National University Hospital, Jongno-gu, Seoul
  - Severance Hospital, Seodaemun-gu, Seoul
  - Asan Medical Center, Songpa-gu, Seoul

REFERENCES:
- [Derived] Kim JY, Park K, Im SA, Jung KH, Sohn J, Lee KS, Kim JH, Yang Y, Park YH. Clinical implications of HER2 mRNA expression and intrinsic subtype in refractory HER2-positive metastatic breast cancer treated with pan-HER inhibitor, poziotinib. Breast Cancer Res Treat. 2020 Dec;184(3):743-753. doi: 10.1007/s10549-020-05891-0. Epub 2020 Aug 28. PMID 32860168